CLINICAL TRIAL: NCT03398616
Title: Regulation of Retinal Blood Flow in Response to an Experimental Increase in Intraocular Pressure
Brief Title: Regulation of Retinal Bloodflow Pressure
Status: Completed | Type: Observational
Sponsor: Gerhard Garhofer (Other)
Responsible Party: Sponsor-Investigator, Gerhard Garhofer, Assoc.Prof.PD, MD, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: OPHT-080515
Record Dates: First submitted 2018-01-08; First posted 2018-01-12 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Retinal Bloodflow
Keywords: Retinal Bloodflow Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Autoregulation is defined as the ability of a vascular bed to adapt its vascular resistance to changes in perfusion pressure. In the eye, several studies have reported that retinal blood flow is autoregulated over a wide range of ocular perfusion pressures. Large scale studies have shown that reduced ocular perfusion pressure is an important risk factor for the prevalence, the incidence and the progression of primary open angle glaucoma. There is also evidence that autoregulation is impaired in patients with primary open angle glaucoma.

To gain more insight into these phenomena in humans is the primary goal of the present study.

The present study aims to investigate the pressure/flow relationship as a measure for retinal blood flow autoregulation during an experimental increase in intraocular pressure by the use of the suction cup technique. Retinal blood flow will be measured by Doppler OCT.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years
* Non-smokers
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropy < 1 Dpt.

Exclusion Criteria:- Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study

* Treatment in the previous 3 weeks with any drug (except contraceptives)
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks
* Pregnancy, planned pregnancy or lactating

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 16 healthy subjects
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Retinal pressure-flow-relationship as assessed with FDOCT | 01.02.2018-31.12.2018

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Puchner S, Schmidl D, Ginner L, Augustin M, Leitgeb R, Szegedi S, Stjepanek K, Hommer N, Kallab M, Werkmeister RM, Schmetterer L, Garhofer G. Changes in Retinal Blood Flow in Response to an Experimental Increase in IOP in Healthy Participants as Assessed With Doppler Optical Coherence Tomography. Invest Ophthalmol Vis Sci. 2020 Feb 7;61(2):33. doi: 10.1167/iovs.61.2.33. PMID 32084274